CLINICAL TRIAL: NCT03046706
Title: Is Voice Rest Contributes to the Quality of Voice After Surgery to Remove Benign Vocal Cord Lesion?
Brief Title: The Role of Vocal Rest After Removal of Benign Lesions From Vocal Cord
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M.P
Record Dates: First submitted 2017-01-29; First posted 2017-02-08 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Vocal Fold Polyp; Vocal Cord Dysfunction
Keywords: voice rest; laryngeal surgery; glottic polyp; glottic cyst
MeSH Terms: conditions — Vocal Cord Dysfunction

STUDY DESIGN:
Intervention Model Description: The research group is the group of patients who do not keep voice rest and talk without restrictions or special instructions after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard voice rest (Active Comparator): This group maintains postoperative voice rest. Namely, absolute voice rest for a week, followed by a week of relative voice rest sound (talking is allowed for 20 minutes a day). post operative voice rest
  Interventions: Behavioral: post operative voice rest
- no voice rest (Experimental): This group has no limitations regarding post operative speech. Members can talk indefinitely after surgery with no special restrictions.
  Interventions: Behavioral: No voice rest

INTERVENTIONS:
Behavioral: post operative voice rest — After surgery, a week of total silence. In the second week after surgery talking is allowed for 20 minutes a day.
  Arms: standard voice rest
Behavioral: No voice rest — No limitations regarding post operative speech. Members can talk indefinitely after surgery with no special restrictions
  Arms: no voice rest

SUMMARY:
The accepted recommendation after removal of vocal cord lesion is voice rest.This recommendation leads to great tension among the patients, loss of working days and need to practice speech therapy.The investigators hypothesize that voice rest after surgery does not affect the quality of the patient's voice. The investigators will divide the patients into 2 groups: the first group will be instructed for a postoperative voice rest and the second group will not. Later the investigators will compare the results and conclude whether voice rest had any significance.

DETAILED DESCRIPTION:
The prevailing view among laryngologists is that voice rest after laryngeal surgery is important to ensure a good recovery of the epithelium and lamina propria layers of the vocal cord. Speaking immediately after surgery leads to the formation of an irregular collagen in large quantities of the vocal cords - namely the creation scar tissue. The scarred vocal cords leads to a decrease in its elasticity, which is reflected in poor speech quality. Although this theory, not many works were published in the literature proving the necessity for voice rest after vocal cord surgery.

Several studies have been recently published which claim that there is no need for vocal rest and stress the importance of a moderate voice effort straight after surgery. This need is based on the idea that early mobilization of tissue after surgery led to the creation of a healthy soft tissue architecture.

The investigators hypothesize that there is no role for vocal rest after surgery to remove benign lesions from the vocal cords.

Patients candidate for laryngeal surgery that include removal of a benign vocal cord lesion will be divided into two groups:

1. Patients instructed for the conventional post operative voice rest, namely absolute voice rest for a week and another week of relative voice rest (speaking is allowed for 20 minutes a day).
2. Patients instructed to speak freely without restrictions after the surgery. those are the study phases: * first visit- preoperative visit.

   * First the investigators prove by fiber optic examination that the patient suffers from the scourge of benign vocal cord lesion. Then the patient gets an explanation of the study, fill a demographic questionnaire. Next the patient fills the VHI (voice handicap index) questionnaire - a questionnaire which assesses the impact of the patient voice by 3 measures:emotional,functional and psychosocial. The questionnaire contains 30 questions. Any question dotted between 0-4 by the patient so that a higher score means more bad sound.
   * Optical fiber testing is performed. Vocal cords including the lesion are photographed and video files are saved . Stroboscopic test for determining the quality of vibration, movement and closure of the vocal cords.The patient voice is recorded for future determination of the GRBAS (Grade,Roughness, breathiness, asthenia,strain). this index, scored by the laryngologists assesses the patient's voice according to five factors- grade, roughness, breathiness, asthenia,strain. Each parameter dotted between 0-3 so a higher score means more bad sound.The last test is objective. The voice recording will undergo computer analysis which determine the following voice objectives : fundamental frequency, jitter, shimmer, harmonic to noise ratio.

Lastly the patient is randomized (by block randomization) to determine to which group the patient belongs.

Patients belonging to the control group (standard post operative voice rest) receive a form where they annotate every day whether they kept on the instructed sound regime. This log will allow the investigators to track the compliance of the patients belonging to the voice rest group.

* Second visit- 3 days post operative

  * Execute an optical fiber examination for description and evaluation of the recovery process of the vocal cord.
  * Vocal cords including the lesion will be photographed and video files are saved. stroboscopic test for future determination of the quality of vibration, movement and closure of the vocal cods.
* Third visit- 14 days post operative

Same examination as the second visit are performed plus:

- The patient voice will be recorded to determine the GRBAS Index by the laryngologist. recording of the patient's voice for an objective voice analysis evaluation using a computer.

* Forth visit- 1 months post operative. Same examinations as the second visit are performed.
* Fifth visit- 3 months post operative. Same examinations as the second visit are performed plus patient fills VHI questionnaire.
* Sixth visit- 6 months post operative. Same examinations as the fifth visit are performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient Over 18 years old suffers a benign vocal cord lesion and candidate for surgical removal . Recruitment will take place in the voice and Swallowing Clinic. Rambam medical center. Israel.

Exclusion Criteria:

* A patient under 18.
* Demented patient.
* Deaf patient.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Patient's evaluation of his own voice | 1 month post operative
  VHI questionnaire score
Patient's evaluation of his own voice | 3 months post operative
  VHI questionnaire score
Patient's evaluation of his own voice | 6 months post operative
  VHI questionnaire score
doctors evaluation of the patient's voice | 1 month post operative
  GRABS scale score
doctors evaluation of the patient's voice | 3 month post operative
  GRABS scale score
doctors evaluation of the patient's voice | 6 month post operative
  GRABS scale score
voice analysis by a software | 1 month post operative
  jitter score, shrimmer score, harmonic to noise ration
voice analysis by a software | 3 month ost operative
  jitter score, shrimmer score, harmonic to noise ration
voice analysis by a software | 6 month post operative
  jitter score, shrimmer score, harmonic to noise ration

SECONDARY OUTCOMES:
Testing the effect of various regimens voice rest on the healing process of vocal cords. the parameters the will be tested are : edema, hyperemia, epithelization, other (presence of granuloma/web) | 3 days post operative
  The next parameters will be evaluated in each visit:
  1. edema- scoring the edema severity .score 1= mild edema .score 2= moderate edema score 3= severe edema hyperemia- scoring the hyperemia severity .score 1= mild hyperemia .score 2= moderate hyperemia score 3= severe hyperemia epithelization degree: 1 =up to 20% 2= up to 50% 3= up to 75% 4- complete epithelization other findings: 1= granuloma 2= web. The final score of each visit includes the sum of all scores separately and will be reported as a single value.
Testing the effect of various regimens voice rest on the healing process of vocal cords. the parameters the will be tested are : edema, hyperemia, epithelization, other (presence of granuloma/web) | 2 weeks post operative
  The next parameters will be evaluated in each visit:
  1. edema- scoring the edema severity .score 1= mild edema .score 2= moderate edema score 3= severe edema hyperemia- scoring the hyperemia severity .score 1= mild hyperemia .score 2= moderate hyperemia score 3= severe hyperemia epithelization degree: 1 =up to 20% 2= up to 50% 3= up to 75% 4- complete epithelization other findings: 1= granuloma 2= web. The final score of each visit includes the sum of all scores separately and will be reported as a single value.
Testing the effect of various regimens voice rest on the healing process of vocal cords. the parameters the will be tested are : edema, hyperemia, epithelization, other (presence of granuloma/web) | 1 month post operative
  The next parameters will be evaluated in each visit:
  1. edema- scoring the edema severity .score 1= mild edema .score 2= moderate edema score 3= severe edema hyperemia- scoring the hyperemia severity .score 1= mild hyperemia .score 2= moderate hyperemia score 3= severe hyperemia epithelization degree: 1 =up to 20% 2= up to 50% 3= up to 75% 4- complete epithelization other findings: 1= granuloma 2= web. The final score of each visit includes the sum of all scores separately and will be reported as a single value.
Testing the effect of various regimens voice rest on the healing process of vocal cords. the parameters the will be tested are : edema, hyperemia, epithelization, other (presence of granuloma/web) | 3 month post operative
  The next parameters will be evaluated in each visit:
  1. edema- scoring the edema severity .score 1= mild edema .score 2= moderate edema score 3= severe edema hyperemia- scoring the hyperemia severity .score 1= mild hyperemia .score 2= moderate hyperemia score 3= severe hyperemia epithelization degree: 1 =up to 20% 2= up to 50% 3= up to 75% 4- complete epithelization other findings: 1= granuloma 2= web. The final score of each visit includes the sum of all scores separately and will be reported as a single value.
Testing the effect of various regimens voice rest on the healing process of vocal cords. the parameters the will be tested are : edema, hyperemia, epithelization, other (presence of granuloma/web) | 6 month post operative
  The next parameters will be evaluated in each visit:
  1. edema- scoring the edema severity .score 1= mild edema .score 2= moderate edema score 3= severe edema hyperemia- scoring the hyperemia severity .score 1= mild hyperemia .score 2= moderate hyperemia score 3= severe hyperemia epithelization degree: 1 =up to 20% 2= up to 50% 3= up to 75% 4- complete epithelization other findings: 1= granuloma 2= web. The final score of each visit includes the sum of all scores separately and will be reported as a single value.

CONTACTS AND LOCATIONS:
Overall Officials: ziv gil, MD, Study Director — Head of ear nose throat department Rambam medical center Israel
Locations (1):
- Rambam medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Behrman A, Sulica L. Voice rest after microlaryngoscopy: current opinion and practice. Laryngoscope. 2003 Dec;113(12):2182-6. doi: 10.1097/00005537-200312000-00026. PMID 14660924
- [Background] Ishikawa K, Thibeault S. Voice rest versus exercise: a review of the literature. J Voice. 2010 Jul;24(4):379-87. doi: 10.1016/j.jvoice.2008.10.011. Epub 2009 Aug 5. PMID 19660903
- [Background] Kiagiadaki D, Remacle M, Lawson G, Bachy V, Van der Vorst S. The effect of voice rest on the outcome of phonosurgery for benign laryngeal lesions: preliminary results of a prospective randomized study. Ann Otol Rhinol Laryngol. 2015 May;124(5):407-12. doi: 10.1177/0003489414560583. Epub 2014 Nov 20. PMID 25416241
- [Background] Rousseau B, Gutmann ML, Mau T, Francis DO, Johnson JP, Novaleski CK, Vinson KN, Garrett CG. Randomized controlled trial of supplemental augmentative and alternative communication versus voice rest alone after phonomicrosurgery. Otolaryngol Head Neck Surg. 2015 Mar;152(3):494-500. doi: 10.1177/0194599814566601. Epub 2015 Jan 20. PMID 25605690
- [Background] Kaneko M, Shiromoto O, Fujiu-Kurachi M, Kishimoto Y, Tateya I, Hirano S. Optimal Duration for Voice Rest After Vocal Fold Surgery: Randomized Controlled Clinical Study. J Voice. 2017 Jan;31(1):97-103. doi: 10.1016/j.jvoice.2016.02.009. Epub 2016 Aug 1. PMID 27492336
- [Background] J. A. Koufman, P.D Blalock. Is voice rest never indicated? J. voice Vol 3, No. 1 87-91